CLINICAL TRIAL: NCT02810808
Title: Random, Open-label Multicenter, Phase IV Study Assessing the Safety and Efficacy of Two Regimens of Ranibizumab 0.5 mg in Chinese Patients With Neovascular AMD
Brief Title: Safety and Efficacy of Two Regimens of Ranibizumab 0.5 mg in Chinese Patients With Neovascular AMD
Acronym: ARTIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other); Shanghai 10th People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor and Executive Vicechair of Department of Ophthalmology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13411950400
Record Dates: First submitted 2014-05-03; First posted 2016-06-23 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular Age-related Macular Degeneration; Ranibizumab; Pro Re Nata
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab 0.5 mg 1+PRN (Experimental): PRN intravitreal injections of ranibizumab 0.5 mg guided by BCVA stabilization in the 11 month treatment period Intervention: Drug: Ranibizumab
  Interventions: Procedure: 1+PRN; Drug: Ranibizumab
- Ranibizumab 0.5 mg 3+PRN (Active Comparator): PRN intravitreal injections of ranibizumab 0.5 mg guided by BCVA stabilization after three Monthly intravitreal injections of the same dose.
  Interventions: Procedure: 3+PRN; Drug: Ranibizumab

INTERVENTIONS:
Procedure: 1+PRN — PRN intravitreal injections of Ranibizumab 0.5mg guided by BCVA stabilization after the injection of the same does at the first month.
  Arms: Ranibizumab 0.5 mg 1+PRN
Procedure: 3+PRN — PRN intravitreal injections of Ranibizumab 0.5mg guided by BCVA stabilization after the first three monthly intravitreal injections of the same does.
  Arms: Ranibizumab 0.5 mg 3+PRN
Drug: Ranibizumab — Ranibizumab - a recombinant, humanized monoclonal antibody Fab that neutralizes all active forms of VEGF-A was recently approved by the Food and Drug Administration for the treatment of all angiographic subtypes of subfoveal neovascular age-related macular degeneration
  Other Names: Lucentis

SUMMARY:
The study will evaluate the efficacy and safety of two different dosing regimens of ranibizumab (0.5 mg on BCVA by 1+PRN vs 3+PRN) in Chinese patients with wet AMD. This study is to provide long-term safety data in the treatment of Chinese patients with wet AMD.

DETAILED DESCRIPTION:
Inclusion Criteria： Age ≥ 50 y/o, nAMD patients（including PCV） Best-corrected visual acuity（BCVA） Exclusion Criteria： Previous anti-VEGF treatment within 3 months History of intraocular surgery within 3 months or arrangement of intraocular surgery in the next 6 months from baseline Active or recent intraocular inflammation in the study eye Primary Endpoint： Improvement in BCVA compared to baseline Other： Central Macular Thickness after Treatment，Numbers of Injections

ELIGIBILITY:
Inclusion Criteria:

* Written informed-consent before any evaluation
* Visual impairment due to active CNV,including predominantly classic CNV,minimally classic CNV,occult CNV with no classic component and PCV.
* 50 years old and older
* Chinese
* For study eye: screening and baseline BCVA scores both should be between 78 and 23 words (including 78 and 23 words) (approximately equals to 20/30-20/320 sneeleen vision chart units) while tested at 4 meters with ETDRS vision chart.

Exclusion Criteria:

* Have Stroke and myocardial infarction within 3 months before screening
* Any active periocular and ocular infection and inflammation (including blepharitis, conjunctivitis, keratitis, scleritis, uveitis, intraocular inflammation) while screening and baseline.
* Uncontrolled glaucoma (under treatment [IOP] ≥ 30 mm Hg or depend on researchers) while screening and baseline
* Neovascularization of iris and neovascular glaucoma while screening and baseline
* Any causes led to choroidal neovascularization except Wet AMD (including ICNV,central serous chorioretinopathy,ocular histoplazmoza and pathologic myopia) while screening and baseline
* With structure injury (including vitreous macular traction,epiretinal membrane involving in central fovea,subretinal fibroplasia,laser scar and central fovea atrophy) within 0.5 optic disc diameter to the central of macula while screening and baseline, which may harm the improvement of vision by treatment according to researchers
* Any systemic anti-VEGF medication(as Avastin) use within 3 months before screening
* Any medication systemic use toxic to lens, retina and optic nerve,including iron amine, chloroquine/chloroquine (Plaquenil ®), tamoxifen, phenothiazine and ethambutol
* For study eye：Used to accept following treatments for wet AMD within 3 months or accept following treatments more than three times before baseline: a)Anti-angiogenesis drugs(pegaptanib （Macugen®），ranibizumab ,bevacizumab（Avastin®),VEGF-Trap，KH902；b）Anecortave acetate corticosteroids；c）Protein kinase C inhibitors，squalamine，siRNA; d)PDT （Visudyne®）treatment,external beam radiotherapy, local laser photocoagulation, vitrectomy, submacular surgery and transpupillary thermotherapy
* Any intraocular surgery(including YAG laser) within 3 months before baseline or predicated within 6 months after baseline
* Intraocular or periocular treatment of corticosteroids within 3 months before baseline
* For follow eye:Any anti-angiogenesis treatment(including anti-VEGF,like Lucentis,Avastin® and KH902 ) within 3 months before baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Mean Snellen BCVA at every visit | 12 months
  Compare of mean Snellen Best-Corrected-visual-acuity and mean central macular thickness by OCT at every visit or treatment between the two groups to assess the efficacy of 1+PRN of Ranibizumab.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 12 months
  Compare of Number of participants with treatment-related adverse events between the two groups to assess the safety of 1+PRN of Ranibizumab.
Mean number of injections in 12 months | 12 months
  Compare of mean number of injection in 12 months between the two groups to assess the efficacy of 1+PRN of Ranibizumab.
mean central macular thickness at every visit by OCT | 12 months
  Compare of mean central macular thickness by OCT at every visit between the two groups to assess the efficacy of 1+PRN of Ranibizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University
Locations (5):
- China (5):
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Shanghai 10th People's Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman DS, Katz J, Bressler NM, Rahmani B, Tielsch JM. Racial differences in the prevalence of age-related macular degeneration: the Baltimore Eye Survey. Ophthalmology. 1999 Jun;106(6):1049-55. doi: 10.1016/S0161-6420(99)90267-1. PMID 10366070
- [Background] Smith W, Assink J, Klein R, Mitchell P, Klaver CC, Klein BE, Hofman A, Jensen S, Wang JJ, de Jong PT. Risk factors for age-related macular degeneration: Pooled findings from three continents. Ophthalmology. 2001 Apr;108(4):697-704. doi: 10.1016/s0161-6420(00)00580-7. PMID 11297486
- [Background] Hsu WM, Cheng CY, Liu JH, Tsai SY, Chou P. Prevalence and causes of visual impairment in an elderly Chinese population in Taiwan: the Shihpai Eye Study. Ophthalmology. 2004 Jan;111(1):62-9. doi: 10.1016/j.ophtha.2003.05.011. PMID 14711715
- [Background] Miyazaki M, Nakamura H, Kubo M, Kiyohara Y, Oshima Y, Ishibashi T, Nose Y. Risk factors for age related maculopathy in a Japanese population: the Hisayama study. Br J Ophthalmol. 2003 Apr;87(4):469-72. doi: 10.1136/bjo.87.4.469. PMID 12642312
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Lalwani GA, Rosenfeld PJ, Fung AE, Dubovy SR, Michels S, Feuer W, Davis JL, Flynn HW Jr, Esquiabro M. A variable-dosing regimen with intravitreal ranibizumab for neovascular age-related macular degeneration: year 2 of the PrONTO Study. Am J Ophthalmol. 2009 Jul;148(1):43-58.e1. doi: 10.1016/j.ajo.2009.01.024. Epub 2009 Apr 18. PMID 19376495
- [Background] Tano Y, Ohji M; EXTEND-I Study Group. EXTEND-I: safety and efficacy of ranibizumab in Japanese patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration. Acta Ophthalmol. 2010 May;88(3):309-16. doi: 10.1111/j.1755-3768.2009.01843.x. Epub 2010 Feb 16. PMID 20163368
- [Background] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Derived] Wang F, Yuan Y, Wang L, Ye X, Zhao J, Shen M, Zhang Q, Xu D, Qin G, Zhang W, Yuan F, Chang Q, Zhao P, Wang F, Sun X. One-Year Outcomes of 1 Dose versus 3 Loading Doses Followed by Pro Re Nata Regimen Using Ranibizumab for Neovascular Age-Related Macular Degeneration: The ARTIS Trial. J Ophthalmol. 2019 Oct 10;2019:7530458. doi: 10.1155/2019/7530458. eCollection 2019. PMID 31687203